CLINICAL TRIAL: NCT04553770
Title: A Phase II, Multicenter, Open-Label Trial to Evaluate the Safety and Efficacy of Trastuzumab Deruxtecan (DS-8201a) With or Without Anastrozole for HER2 Low Hormone Receptor Positive (HR+) Breast Cancer in the Neoadjuvant Setting
Brief Title: Trastuzumab Deruxtecan Alone or in Combination With Anastrozole for the Treatment of Early Stage HER2 Low, Hormone Receptor Positive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Translational Research in Oncology-U.S (Unknown); Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-001275; NCI-2020-06086 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Early-stage Breast Cancer; Hormone Receptor Positive Breast Carcinoma; Invasive Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (trastuzumab deruxtecan) (Active Comparator): Patients receive trastuzumab deruxtecan IV over 90 minutes on cycle 1 day 1 and 30 minutes on day 1 of each subsequent cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Interventions: Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab Deruxtecan
- Arm B (trastuzumab deruxtecan, anastrozole) (Experimental): Patients receive trastuzumab deruxtecan IV over 90 minutes on cycle 1 day 1 and 30 minutes on day 1 of each subsequent cycle and anastrozole PO QD on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  Interventions: Drug: Anastrozole; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
  Arms: Arm B (trastuzumab deruxtecan, anastrozole)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; WHO 10516

SUMMARY:
This phase II trial investigates how well trastuzumab deruxtecan works alone or in combination with anastrozole in treating patients with HER2 low, hormone receptor positive breast cancer. Trastuzumab deruxtecan is a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug called deruxtecan. Trastuzumab attaches to HER2 expressed at low levels on cancer cells in a targeted way and delivers deruxtecan to kill them. Anastrozole works by decreasing estrogen production and suppressing the growth of tumors that need estrogen to grow. This study is evaluating how effective trastuzumab deruxtecan is at treating hormone receptor positive cancer cells that have low levels of HER2 expressed on them when given alone or in combination with anastrozole.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify treatment arm with strongest signal of efficacy, based on pathologic complete response (pCR) rate, between two neoadjuvant systemic therapy regimens in participants with early stage, HER2 low, hormone receptor positive (HR+) breast cancer.

SECONDARY OBJECTIVES:

I. To assess the safety profile of the two novel neoadjuvant experimental arms. II. To assess the molecular changes in tumor biomarkers including Ki67 after 1 cycle of targeted therapy.

III. Pathological Assessment According to Residual Cancer Burden (RCB) Index at surgery.

IV. To investigate potential serum and tumor predictive biomarkers to predict response to experimental therapy.

EXPLORATORY OBJECTIVES:

I. To investigate potential serum and tumor predictive biomarkers to predict response to experimental therapy.

II. To assess quality of life by evaluating toxicity burden using a quality of life (QOL)/patient reported outcomes (PRO) questionnaire- the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 (EORTC QLQ-C30) instrument.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive trastuzumab deruxtecan intravenously (IV) over 90 minutes on cycle 1 day 1 and 30 minutes on day 1 of each subsequent cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

ARM B: Patients receive trastuzumab deruxtecan IV over 90 minutes on cycle 1 day 1 and 30 minutes on day 1 of each subsequent cycle and anastrozole orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

After completion of study treatment, patients are followed up at 21-28 days.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated operable invasive carcinoma of the breast greater than 2.0 cm (cT2) in size based on physical exam or imaging. Patients with clinical node negative disease or clinical node (cN1/cN2) positive are allowed provided they are deemed to have operable disease at study entry
* Participants with clinically involved lymph nodes should not have radiological evidence of distant disease per standard of care staging prior to patient informed consent form (PICF) signature
* In the United States
* Tumor is HER2-low by immunohistochemistry (IHC), defined as 1+ or 2+, confirmed by central testing (central testing results not required for enrollment, unless no local results available). If HER2 is 2+ by IHC, fluorescence in situ hybridization (FISH) must be performed (per standard of care) and the FISH result must be HER2 non-amplified per 2018 American Society of Clinical Oncology College of American Pathologists (ASCO CAP) guidelines
* Tumor is HR positive (HR+) per ASCO CAP guidelines with known estrogen and progesterone receptor status, locally defined
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Normal cardiac function (left ventricular ejection fraction [LVEF] >= 50%) based on echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before randomization/enrollment
* Platelet count >= 100 000/mm^3 (Platelet transfusion is not allowed within 1 week prior to screening assessment) (within 14 days before randomization/enrollment)
* Hemoglobin >= 9.0 g/dL (red blood cell transfusion is not allowed within 1 week prior to screening assessment) (within 14 days before randomization/enrollment)
* Absolute neutrophil count (ANC) >=1500/mm^3 (Granulocyte colony-stimulating factor (G-CSF) administration is not allowed within 1 week prior to screening assessment) (within 14 days before randomization/enrollment)
* Creatinine clearance >= 30 mL/min as calculated using the Cockcroft-Gault equation or serum creatinine =< 1.5 x upper limit of normal (ULN) (within 14 days before randomization/enrollment)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) =< 3 x ULN (within 14 days before randomization/enrollment)
* Total bilirubin =< 1.5 x ULN (within 14 days of randomization/enrollment). Participants with Gilbert's syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted
* Serum albumin >= 2.5 g/dL (within 14 days before randomization/enrollment)
* International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (within 14 days before randomization/enrollment)
* Has adequate treatment washout period before randomization/enrollment, defined as:

  * Major surgery >= 4 weeks
  * Chloroquine/hydroxychloroquine > 14 days
* Negative pregnancy test (serum) for women of child bearing potential (CBP):

  * Women are considered of CBP unless: they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment she is considered not of CBP
* Male and female participants of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking trial treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male partner sterilization (at least 6 months prior to randomization). For female patients on the trial the vasectomized male partner should be the sole partner for that patient. If vasectomy of the male partner is the highly effective method of contraception chosen, the success of the vasectomy should be medically confirmed according to local practice
  * Placement of an intrauterine device (IUD)
* Male participants must not freeze or donate sperm starting at screening and throughout the study period, and at least 4 months after the final study drug administration. Preservation of sperm should be considered prior to enrollment in this study
* Female participants must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration
* Estradiol level must be in post-menopausal range per local lab interpretation prior to baseline biopsy

  * Postmenopausal status is defined as:

    * Patient underwent bilateral oophorectomy, or
    * Age >= 60 years, or
    * Age < 60 years and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene or ovarian suppression) and follicle-stimulating hormone (FSH) and plasma estradiol are in the postmenopausal ranges per local normal ranges
  * Note: for women with therapy-induced amenorrhea, serial measurements of FSH and/or estradiol per local clinical guidelines are required for determination of postmenopausal status. All women who do not meet the criteria for postmenopausal status are considered premenopausal for the purpose of this trial
* Pre- or peri-menopausal and amenable to being treated with ovarian function suppression drugs (goserelin, leuprolide, or triptorelin) per standard of care. Patients must have started treatment with ovarian function suppression at least 28 days prior to first dose of study treatment

Exclusion Criteria:

* Recurrent or metastatic breast cancer
* Bilateral breast cancer (multifocal or multicentric breast cancer is allowed provided that all biopsied lesions are HER2 1+ or 2+, not FISH amplified and are HR positive per ASCO guidelines)
* Inflammatory breast cancer
* Prior systemic therapy for invasive cancer

  * Prior tamoxifen for history of ductal breast carcinoma in situ (DCIS) allowed, but no prior aromatase inhibitor, no prior chemotherapy and no prior HER2-targeted therapy
* Prior ipsilateral chest wall radiation
* Major surgery < 4 weeks prior to enrollment
* Medical history of myocardial infarction within 6 months before randomization/enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), troponin levels consistent with myocardial infarction as defined according to the manufacturer 28 days prior to randomization
* Unable to swallow oral medications
* Is pregnant or lactating, or planning to become pregnant
* Corrected QT interval prolongation to > 470 ms (females) or > 450 ms (males) based on average of the screening triplicate 12-lead electrocardiogram
* Known hypercoaguable disorder requiring use of anticoagulant
* Significant gastrointestinal disorders limiting absorption or tolerance of oral medications (for example, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea)
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Has multiple primary malignancies within 3 years, except:

  * Adequately resected non-melanoma skin cancer
  * Curatively treated non breast in-situ disease, and other solid non-breast tumors curatively treated are allowed if > 3 years from diagnosis and no evidence of recurrence in that time
  * Prior history of DCIS is allowed as long as patient has not received an aromatase inhibitor, has not received ipsilateral breast/chest radiation
  * Prior history of contralateral invasive breast cancer (diagnosed by biopsy > 2 years prior to current diagnosis) is allowed provided patient has not received prior aromatase inhibitor, CDK4/6 inhibitor (CDK4/6i), HER2-targeted therapy or chemotherapy and has not experienced any recurrence and has no evidence of recurrence (based on standard clinical evaluation)
* Other concurrent anti-cancer therapy. Note: ovarian function suppression drugs (goserelin, leuprolide, or triptorelin) and/or bone modifying agents (bisphosphonates, denosumab) do not count as anti-cancer therapy for this criteria. If taking bisphosphonates or denosumab, must have been on these agents prior to signing consent
* Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results
* Has known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA). Subjects should be tested for HIV prior to randomization/enrollment if required by local regulations or Institutional Review Board (IRB)/ethics committee (EC)
* Have personal history within the last 12 months of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest
* Have received an autologous or allogeneic stem-cell transplant
* Has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]). Screening is not required for enrollment
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment must be stopped prior to first baseline biopsy
* Has history of severe hypersensitivity reactions to other monoclonal antibodies and/or to either the drug substances or inactive ingredients in the drug product
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (i.e. rheumatoid arthritis, Sjogren's, sarcoidosis etc.), or prior pneumonectomy
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | Baseline to surgery
  pCR is defined as the absence of invasive cancer in the breast and sampled regional lymph nodes. pCR will be calculated along with the corresponding exact 95% Clopper-Pearson confidence interval (CI).

SECONDARY OUTCOMES:
Incidence of adverse events | Starting cycle 1 day 1 (each cycle is 21 days), through study completion, an average of 6 months.
  Overall exposure to study drug, the numbers of participants completing each cycle, and the dose intensity will be summarized using descriptive statistics. The number of participants with any dose adjustment will be presented for entire treatment period as well as for each cycle. The number of participants with dose reductions, dose delays, or dose omissions will also be summarized, as will the reasons for dose adjustments. Adverse events and serious adverse events will be reported using a Common Terminology Criteria for Adverse Events version 5.0 terminology and severity.
Molecular changes in tumor biomarkers including Ki67 expression | Baseline to surgery
  Percent change in Ki67 expression from baseline to the core biopsy obtained between cycle 1 day 17 and cycle 1 day 21, and surgery.
Clinical objective response | Baseline to surgery
  Clinical objective response rate will be estimated and 95% exact Clopper-Pearson CIs will be provided.
Biomarker analyses | Baseline to surgery
  Gene expression and biomarker assay results are exploratory and will be summarized (e.g. mean change in from baseline to during treatment and to prior to surgery) and correlated with clinical outcomes as appropriate.

OTHER OUTCOMES:
Quality of life assessment: questionnaire | Baseline, day 1 of each cycle (each cycle is 21 days) , at study completion, an average of 6 months.
  Will assess quality of life by evaluating toxicity burden using a quality of life/patient reported outcome questionnaire- the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas P McAndrew, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (9):
- United States (9):
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Cancer Blood and Specialty Clinic, Los Alamitos, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Torrance Memorial Physician Network / Cancer Care, Torrance, California
  - PIH Health, Whittier, California
  - Orlando Health, Inc. d/b/a Orlando Health UF Health Center, Orlando, Florida
  - Ft. Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts